CLINICAL TRIAL: NCT01676545
Title: Genetics of Periodontal Diseases in Chinese
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Stomatological Disease Center (Other)
Collaborators: Interleukin Genetics, Inc. (Industry)
Other Study IDs: ILI-10-122-PST2China
Record Dates: First submitted 2012-08-30; First posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Chronic Periodontitis
- Control

SUMMARY:
(A retrospective case control study to validate the association between Interleukin-1 gene variations and adult chronic periodontal disease in Chinese (Shanghai))

ELIGIBILITY:
Inclusion Criteria:

- To be included in this study, an individual needs to be Han Chinese of 35 years of age or older at time of enrollment.

Exclusion Criteria:

- 1) Age younger than 35 years old. 2) Patients with diagnosis of rheumatoid arthritis, psoriasis, inflammatory bowel disease, glomerulonephritis/kidney disease, cancer, or Sjogren's syndrome.

3) Organ transplant recipients.

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All study subjects will be selected from a pre-existing patient database in Shanghai. All chronic periodontitis cases and controls will be subjects who were at least 35 years old at time of enrollment.
  Classification of chronic periodontitis will be based on the extent of periodontal tissue destruction with consideration of tooth loss.
Sampling Method: Non-Probability Sample
Dates: Start 2011-07